CLINICAL TRIAL: NCT01835678
Title: Effects of Linagliptin on Renal Endothelium Function in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRC2012LINA; 2012-002278-30 (EudraCT Number)
Record Dates: First submitted 2013-03-18; First posted 2013-04-19 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Type 2-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin (Active Comparator): Linagliptin
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin — orally 5 mg/d for 4 weeks
  Arms: Linagliptin
Drug: Placebo — orally once a day for 4 weeks
  Arms: Placebo

SUMMARY:
Diabetes mellitus is a metabolic disease with a growing prevalence worldwide, affecting 171 million people in 2000 and an expected 366 million people in 2030 (1) and therefore diabetic nephropathy is rapidly increasing in the Western hemisphere and represents in up to 50 % the cause of end stage renal disease. Hence, early intervention is desirable to prevent any damage to the kidneys. In the early stage of diabetic nephropathy, endothelium dysfunction is a key pathogenetic process as indicated by increased leakage of albumin through the glomerular barrier (2).

Hence, improvement of endothelium function is an attractive therapeutic goal of antidiabetic medication. Endothelial dysfunction, in particular basal nitric oxide activity, has been also identified as pivotal determinant of glomerular filtration rate (3).

A new and promising class of antidiabetic drugs are the gliptins. Gliptins act by inhibiting the enzyme dipeptidyl peptidase-4 (DPP-4), which is responsible for the rapid inactivation of glucagon-like peptide-1 (GLP-1) - an incretin hormone of the gut (6 - 8), thereby enhancing and prolonging the effects of GLP-1. GLP-1 - member of the incretin hormones - is released into the blood after meal ingestion and stimulates the insulin secretion in a glucose dependent manner. This accounts for the marked prandial insulin response, which prevents prandial hyperglycemia.

Apart from surrogate parameters like reduction of fasting and postprandial blood glucose levels or improvement of HbA1c, the effect of gliptins on micro- and macrovascular function and cardiovascular outcome has not been the primary focus of current studies. However, infusion of GLP-1, the incretin hormone affected by gliptins has been reported to ameliorate endothelial dysfunction in patients suffering from coronary artery disease (9) and it was recently shown that infusion of GLP-1 into healthy human subjects increases both normal and ACh-induced vasodilatation (10). In studies on rats with diabetes, GLP-1 infusion nearly re-established their normal vascular tone (11) and there are further data from experimental animals that indicate a beneficial effect of GLP-1 on endothelial function (12).

It is of major interest whether therapy with gliptins improves endothelial function of the micro- and macrovasculature. In face of the burden that diabetic nephropathy causes, the effect of linagliptin on the renal vasculature and endothelium integrity of the renal circulation (as measured by the availability of nitric oxide), is a key stone in order to claim that linagliptin is an effective antidiabetic agents. There is a need to demonstrate that linagliptin is effective beyond its blood glucose lowering actions and improves vascular endothelium function in the kidney.

DETAILED DESCRIPTION:
Diabetes mellitus is a metabolic disease with a growing prevalence worldwide, affecting 171 million people in 2000 and an expected 366 million people in 2030 (1) and therefore diabetic nephropathy is rapidly increasing in the Western hemisphere and represents in up to 50 % the cause of end stage renal disease. Hence, early intervention is desirable to prevent any damage to the kidneys. In the early stage of diabetic nephropathy, endothelium dysfunction is a key pathogenetic process as indicated by increased leakage of albumin through the glomerular barrier (2).

Hence, improvement of endothelium function is an attractive therapeutic goal of antidiabetic medication. Endothelial dysfunction, in particular basal nitric oxide activity, has been also identified as pivotal determinant of glomerular filtration rate (3). Previously, blockade of the renin angiotensin system have been found to be effective in improving endothelium function (4). Furthermore, we observed that renal endothelium function is improved by cardiovascular risk factor control (e.g. blood pressure) and may be predictive for the development of diabetic nephropathy (5).

A new and promising class of antidiabetic drugs are the gliptins. Gliptins act by inhibiting the enzyme dipeptidyl peptidase-4 (DPP-4), which is responsible for the rapid inactivation of glucagon-like peptide-1 (GLP-1) - an incretin hormone of the gut (6 - 8), thereby enhancing and prolonging the effects of GLP-1. GLP-1 - member of the incretin hormones - is released into the blood after meal ingestion and stimulates the insulin secretion in a glucose dependent manner. This accounts for the marked prandial insulin response, which prevents prandial hyperglycemia. Several efficacy studies demonstrated a significant improvement of HbA1c with gliptins. In addition, gliptins improved fasting as well as prandial glucose levels and did not induce weight gain. Due to these positive metabolic effects in combination with a very small spectrum of side effects gliptins might very well be part of the standard therapy for type 2 diabetes in the future.

Apart from surrogate parameters like reduction of fasting and postprandial blood glucose levels or improvement of HbA1c, the effect of gliptins on micro- and macrovascular function and cardiovascular outcome has not been the primary focus of current studies. However, infusion of GLP-1, the incretin hormone affected by gliptins has been reported to ameliorate endothelial dysfunction in patients suffering from coronary artery disease (9) and it was recently shown that infusion of GLP-1 into healthy human subjects increases both normal and ACh-induced vasodilatation (10). In studies on rats with diabetes, GLP-1 infusion nearly re-established their normal vascular tone (11) and there are further data from experimental animals that indicate a beneficial effect of GLP-1 on endothelial function (12).

Diabetes mellitus is strongly associated with microangiopathy and macroangiopathy and is a strong independent risk factor for cardiovascular disease and cardiovascular mortality (13). Endothelial dysfunction which plays a crucial role in the atherosclerotic process is commonly observed in patients with diabetes mellitus and already prediabetes and has - amongst other factors - been linked to fasting and postprandial hyperglycemia. Gliptins reduce hyperglycemia and hyperglycemic peaks by preventing inactivation of GLP-1, which exerted beneficial effects on the endothelium in previous studies.

It is of major interest whether therapy with gliptins improves endothelial function of the micro- and macrovasculature. In face of the burden that diabetic nephropathy causes, the effect of linagliptin on the renal vasculature and endothelium integrity of the renal circulation (as measured by the availability of nitric oxide), is a key stone in order to claim that linagliptin is an effective antidiabetic agents. There is a need to demonstrate that linagliptin is effective beyond its blood glucose lowering actions and improves vascular endothelium function in the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged between 18 and 70 years
* Type 2 diabetes without diabetic nephropathy (definition see exclusion criteria)

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Use of insulin, glitazone or gliptins within the past 3 months
* Any other oral antidiabetic drug that can not be discontinued for the study period.
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 6 months prior to study inclusion
* Urinary albumin excretion (UACR) > 100 mg/g (early morning spot urine)
* eGFR <45 ml/min/1.73m² (MDRD Formula)
* Uncontrolled arterial hypertension (RR ≥180/ ≥110mmHg)
* HbA1c ≥ 10%
* Fasting plasma glucose ≥ 240 mg/dl
* Body mass index ≥ 40 kg/m²
* Triglyceride levels ≥ 1000 mg/dl
* HDL-cholesterol levels <25 mg/dl
* Overt congestive heart failure (CHF) or history of CHF
* Severe disorders of the gastrointestinal tract or other diseases which interfere the pharmacodynamics and pharmacokinetics of study drugs
* Significant laboratory abnormalities such as SGOT or SGPT levels more than 3 x above the upper limit of normal range, serum creatinine > 2mg/dl
* Drug or alcohol abuses
* Pregnant or breast-feeding patients
* Any patient currently receiving chronic (>30 consecutive days) treatment with an oral corticosteroid
* Patients being treated for severe auto immune disease e.g. lupus
* Participation in another clinical study within 30 days prior to visit 1
* Individuals at risk for poor protocol or medication compliance
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
effect of linagliptin compared to placebo on basal production and release of nitric oxide (NO) from renal vasculature | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  The primary objective of the study is the change of renal plasma flow to LNMMA infusion from baseline (given in ml/min) to determine the effect of linagliptin compared to placebo on basal production and release of nitric oxide (NO) from renal vasculature.

SECONDARY OUTCOMES:
effects of linagliptin compared to placebo on other renal hemodynamic parameters | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  Renal plasma flow, glomerular filtration rate and filtration fraction, renal vascular resistance, calculated intraglomerular pressure.
effect of linagliptin compared to placebo on urinary albumin creatinine ratio and tubular markers (e.g. NGAL). | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  effect of linagliptin compared to placebo on urinary albumin creatinine ratio and tubular markers (e.g. NGAL).
effect of linagliptin compared to placebo on markers of oxidative stress (e.g. isoprostanes) and inflammation (e.g. hsCRP). | Changes from baseline after 4 weeks with linagliptin versus placebo
  effect of linagliptin compared to placebo on markers of oxidative stress (e.g. isoprostanes) and inflammation (e.g. hsCRP).
effect of linagliptin compared to placebo on metabolic parameters (fasting glucose, fasting insulin, triglycerides, total-, LDL- and HDL-cholesterol) | Changes from baseline after 4 weeks of treatment with linaplitpin and placebo
  effect of linagliptin compared to placebo on metabolic parameters (fasting glucose, fasting insulin, triglycerides, total-, LDL- and HDL-cholesterol)
effect of linagliptin compared to baseline on the change of renal plasma flow due to L-NMMA-infusion | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  effect of linagliptin compared to baseline on the change of renal plasma flow due to L-NMMA-infusion
effects of linagliptin compared to baseline on other renal hemodynamic parameters | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  effects of linagliptin compared to baseline on other renal hemodynamic parameters: Renal plasma flow, glomerular filtration rate and filtration fraction, renal vascular resistance, calculated intraglomerular pressure
of linagliptin compared to baseline on urinary albumin creatinine ratio and tubular markers (e.g. NGAL) | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  of linagliptin compared to baseline on urinary albumin creatinine ratio and tubular markers (e.g. NGAL)
effect of linagliptin compared to baseline on markers of oxidative stress (e.g. isoprostanes) and inflammation (e.g. hsCRP). | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  effect of linagliptin compared to baseline on markers of oxidative stress (e.g. isoprostanes) and inflammation (e.g. hsCRP)
effect of linagliptin compared to baseline on metabolic parameters (fasting glucose, fasting insulin, triglycerides, total-, LDL- and HDL-cholesterol) | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  effect of linagliptin compared to baseline on metabolic parameters (fasting glucose, fasting insulin, triglycerides, total-, LDL- and HDL-cholesterol)
determine the relationship between changes of renal endothelial function with metabolic changes and changes of isoprostanes | Changes from baseline after 4 weeks of treatment with linagliptin and placebo
  determine the relationship between changes of renal endothelial function with metabolic changes and changes of isoprostanes

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (2):
- Germany (2):
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Nuremberg

REFERENCES:
- [Background] Ott C, Schneider MP, Delles C, Schlaich MP, Schmieder RE. Reduction in basal nitric oxide activity causes albuminuria. Diabetes. 2011 Feb;60(2):572-6. doi: 10.2337/db09-1630. PMID 21270268
- [Background] Schlaich MP, Schmitt D, Ott C, Schmidt BM, Schmieder RE. Basal nitric oxide synthase activity is a major determinant of glomerular haemodynamics in humans. J Hypertens. 2008 Jan;26(1):110-6. doi: 10.1097/HJH.0b013e3282f1a93e. PMID 18090547
- [Background] Ritt M, Ott C, Raff U, Schneider MP, Schuster I, Hilgers KF, Schlaich MP, Schmieder RE. Renal vascular endothelial function in hypertensive patients with type 2 diabetes mellitus. Am J Kidney Dis. 2009 Feb;53(2):281-9. doi: 10.1053/j.ajkd.2008.10.041. Epub 2008 Dec 19. PMID 19100670
- [Result] Ott C, Kistner I, Keller M, Friedrich S, Willam C, Bramlage P, Schmieder RE. Effects of linagliptin on renal endothelial function in patients with type 2 diabetes: a randomised clinical trial. Diabetologia. 2016 Dec;59(12):2579-2587. doi: 10.1007/s00125-016-4083-4. Epub 2016 Sep 1. PMID 27586249